CLINICAL TRIAL: NCT01366859
Title: Nutritional Intervention Using Supplementation With Cysteine-Rich Whey Protein Isolate (Immunocal®) in Children With Autism: Effects in Core Areas of Behavior- A Randomized Double-Blind Study
Brief Title: Nutritional Intervention in Children With Autism Using Whey Protein (Immunocal): Impact on Core Areas of Behavior
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: Immunotec Inc. (Industry)
Responsible Party: Principal Investigator, Ana Maria Castejon Ph.D., Associate Professor, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 01291001F
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-03

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism; Children; Behavior; Glutathione; Whey Protein; Immunocal; Antioxidant
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Behavior | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whey Protein (Immunocal®) (Experimental): The experimental study group will consist of thirty children that will be treated with Immunocal® 0.5 g/kg if less than 18 kg of body weight or 10 g/day for those children over 18 kg of body weight for three months.
  Interventions: Dietary Supplement: Whey Protein
- Placebo: Rice Protein (Placebo Comparator): The control or placebo study arm will consist of thirty children who will receive a dose of 0.5 g/kg of weight a day up to 18 kg of weight a day or a dose of 10 g/day for those over 18 kg for three months.
  Interventions: Dietary Supplement: Rice Protein (Placebo)

INTERVENTIONS:
Dietary Supplement: Whey Protein — The experimental study group will consist of thirty children that will be treated with Immunocal® 0.5 g/kg if less than 18 kg of body weight or 10 g/day for those children over 18 kg of body weight for three months to determine the supplement's effect in core areas of behavior in children with autism.
  Other Names: Immunocal; Cystine-rich Whey Protein Isolate
  Arms: Whey Protein (Immunocal®)
Dietary Supplement: Rice Protein (Placebo) — The control or placebo study group will consist of thirty children that will be treated with rice protein (placebo) 0.5 g/kg if less than 18 kg of body weight or 10 g/day for those children over 18 kg of body weight for three months.
  Arms: Placebo: Rice Protein

SUMMARY:
This study will evaluate the effects of a cysteine-rich whey protein isolate supplement (Immunocal®) on autistic behavior in pre-school children with autism.

DETAILED DESCRIPTION:
Summary:

Autism is a neurodevelopmental disorder currently affecting as many as 1 of 150 children in the United States. Autism is considered by many to be a permanent condition with little hope for improvement. The treatment for autism is centered on special schooling and behavioral therapy; and conventional medical treatments have had little impact on ameliorating this disorder. Recent research has discovered that some autistic individuals have increased markers of oxidative stress and some degree of mitochondrial dysfunction. Furthermore, genetic abnormalities in the glutathione pathway have been associated to autism. Thus, we are proposing that a nutritional supplement based on bovine milk serum containing cysteine-rich whey proteins serving as glutathione precursors can improve behavioral function in children with Autism.

Hypothesis:

Many children with autism have impaired antioxidant/detoxification capacity and chronic oxidative stress. Studies have also shown that autistic children show an abnormally high prevalence of glutathione deficiency. A cysteine-rich whey protein supplement demonstrated to raise glutathione levels will improve the metabolic imbalance and improve measures of autistic behavior.

Purpose:

This study will evaluate the effects of a cysteine-rich whey protein isolate supplement (Immunocal®) on autistic behavior in pre-school children with autism.

Methods:

This will be a 3 month double-blind placebo-controlled study. A total of 60 subjects will be selected/recruited and enrolled (see inclusion and exclusion criteria) to have a minimum 40 evaluable children (including estimated drop-outs) ranging in age from 3 to 5 years old to participate in the study and data recorded and collected. Children will be randomly assigned to either treatment- to the study product (Immunocal) or to the control (rice protein) for three months (20 subjects per group). Core areas of autistic behavior that will be assessed before (baseline/week 0), and at the end of treatment (week 12) are: atypical autistic behaviors and severity, communication, developmental status and behavioral problems. In addition, blood glutathione levels will be quantified before and after treatment. Side effects and adverse reactions will be compared between the two groups before (baseline/week 0) and at the end of treatment (week 12).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV)
* Male/female
* Aged 3-5 years

Exclusion Criteria:

* Milk Allergy
* Rice allergy
* Nut Allergy
* Major medical problems including cardiac, liver endocrine or renal disease
* History of seizure disorder or gross neurological deficit
* Concomitant treatment with psychiatric medication
* Current diet supplementation with N-acetyl-cysteine, alpha lipoic acid or whey protein.
* Comorbid diagnosis: Fragile X syndrome, tuberous sclerosis, phenylketonuria or fetal alcohol syndrome
* Acute illness

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2011-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Behavioral Analysis | Outcome measure assessed at baseline (week 0) and week 12.
  Behavioral analysis will be performed in areas of autism behaviors and severity, communication, developmental status and behavioral problems to establish the effects of a 90 day diet supplementation with a cysteine-rich whey protein isolate (Immunocal®) on autistic behavior in children with a diagnosis of autism according to DSM-IV,

SECONDARY OUTCOMES:
Safety Analysis | Outcome measure assessed at baseline (week 0) and week 12.
  Safety analyses will be conducted to identify any adverse event during the course of the study, doing so will verify the tolerability of a cysteine-rich whey protein supplement (Immunocal®) in children with autism.
Intracellular Glutathione & Antioxidant Capacity | Outcome measured at baseline (week 0) and week 12.
  Reduced and oxidized Glutathione levels in white blood cells will be quantified and correlated with behavioral changes in children with autism supplemented with a cysteine-rich whey protein.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Maria Castejon, Ph.D., Principal Investigator — College of Pharmacy, Nova Southeastern University
Locations (3):
- United States (3):
  - Mailman Segal Center, Fort Lauderdale, Florida
  - Nova Southeastern University Clinic, Fort Lauderdale, Florida
  - Nova Southeastern University, College of Pharmacy, Fort Lauderdale, Florida

REFERENCES:
- [Derived] Castejon AM, Spaw JA, Rozenfeld I, Sheinberg N, Kabot S, Shaw A, Hardigan P, Faillace R, Packer EE. Improving Antioxidant Capacity in Children With Autism: A Randomized, Double-Blind Controlled Study With Cysteine-Rich Whey Protein. Front Psychiatry. 2021 Sep 30;12:669089. doi: 10.3389/fpsyt.2021.669089. eCollection 2021. PMID 34658941